CLINICAL TRIAL: NCT07159568
Title: Visits by Pet Dogs to Patients Admitted to Intensive Care at the Clermont-Ferrand University Hospital: Feasibility Study
Brief Title: Pets Enhancing Therapeutics in Intensive Care Units
Acronym: PET-ICU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AOI 2024 LALANDE; 2025-A00615-44 (Other: ANSM)
Record Dates: First submitted 2025-08-27; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: Intensive Care Unit (ICU) Patients; Dog Therapy
Keywords: dog therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pet dog visit (Experimental)
  Interventions: Other: Pet dog visit

INTERVENTIONS:
Other: Pet dog visit — Pet dog visit will take place during dedicated time slots, following prior verification of the dog's hygiene criteria. The dog may stay in the patient's room for a maximum of 15 minutes. After the visit, an evaluation questionnaire will be completed by the healthcare staff and by the relative who accompanied the dog. The patient's evaluation questionnaire will be completed at ICU discharge if patient is able to respond, or at most 28 days after inclusion if the patient remains in the ICU.

SUMMARY:
Intensive Care Units (ICUs) are well known for their therapeutic and environmental aggressiveness. Current recommendations for the management of critically ill patients, including the "ABCDEF bundle," emphasize family engagement and liberal visitation policies for relatives and loved ones, with the aim of improving patient well-being during their ICU stay.

In France, half of all households own a pet. This close relationship between humans and animals explains why animals have long been involved in medical care. The earliest known use of animals in medicine dates back to the 9th century in Belgium, where they were used to assist individuals with mental illness. More recently, companion animal-assisted interventions have attracted growing interest due to their potential diagnostic and/or therapeutic value, as they may enhance the patient experience during hospitalization. The feasibility, safety, and potential benefits of pet visitation policies have mainly been assessed in conventional hospital wards, but remain understudied in the ICU setting. In France, to our knowledge, only three hospitals have allowed pet visits in the ICU, and these occurred outside of any research protocol.

The study primary objective is to assess the feasibility of companion dog visits in three medical-surgical ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 years or older,
* Admitted to one of the participating ICUs at Clermont-Ferrand University Hospital (Estaing Adult ICU, Montpied Medical-Surgical ICU, or Montpied Neuro-ICU) with an expected ICU stay of 48 hours or more,
* Owner of a companion dog, with family members or relatives able to bring the dog to the ICU.

Exclusion Criteria:

Patient-related exclusion criteria:

* Refusal by the patient or by their family/relatives to participate,
* Lack of affiliation with the French national health insurance system (Sécurité Sociale),
* Patient deprived of liberty or under legal protection (guardianship, curatorship, or judicial safeguard),
* Pregnant or breastfeeding patient,
* Agitated patient, defined as a Richmond Agitation-Sedation Scale (RASS) score > 0 (monitored every four hours according to current standard practice),
* Patient with immunosuppression, defined as: blood neutrophil count < 0.5 G/L, ongoing or recent (within the past month) treatment for solid or hematologic cancer (e.g., chemotherapy, radiotherapy, cell therapy), or receiving immunosuppressive drugs (including organ transplant recipients or corticosteroid therapy for more than two weeks),
* Patient with known colonization by multidrug-resistant bacteria (as routinely assessed upon ICU admission and weekly thereafter),
* Patient with one or more open wounds or injuries that cannot be covered with a dressing.

Dog-related exclusion criteria:

* Dog belonging to category 1 or 2 breeds considered dangerous under current French regulations,
* Dog that never leaves the home environment,
* Dog with an incomplete vaccination status,
* Dog with a known transmissible disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Success of the pet dog visit | Immediately after the intervention
  The success of the pet dog visit is defined as the entry of the animal into the patient's ICU room under the conditions specified in the study protocol

SECONDARY OUTCOMES:
Patient-related safety events regarding inconvenience or harm | Immediately after the intervention
  Any inconvenience or harm to the patient, regardless of nature (including accidental dislodgement or removal of medical equipment/devices such as tracheal tubes, catheters, drains, etc.)
Patient-related safety events regarding infections | ICU discharge (within a maximum of 28 days)
  New colonization with multidrug-resistant organisms (as assessed upon ICU admission and weekly thereafter); and new ICU-associated infections (as routinely screened according to standard care)
Dog-related events regarding aggression or behavioral issues | Immediately after the intervention
  Any display of aggression or behavioral issues (as defined by the participating veterinarian, e.g., stupor, withdrawal, uncontrolled barking, urination or defecation) during the ICU visit, regardless of whether the dog ultimately entered the patient's room.
Staff-related events regarding inconvenience or harm | Immediately after the intervention
  Any inconvenience or harm to a member of the healthcare team, regardless of nature (e.g., injury, hygiene issues, noise, or behavioral disturbance) during the ICU visit, regardless of whether the dog ultimately entered the patient's room.
Visit conditions in the case of success (excluding the safety criteria listed above) | Immediately after the intervention
  Precise duration of the visit in the patient's room (maximum of 15 minutes, as per protocol), any direct contact between the patient and the dog, and the nature of such interaction.
Reasons for potential visit failure (defined as the inability to bring the animal into the patient's ICU room) | Immediately before the intervention
  Reasons are defined as :
  * Non-compliance with local hygiene guidelines and pre-/intra-visit checklists, as developed specifically for this protocol in collaboration with the hospital's infection control team (CLIN).
  * Non-compliance with local veterinary regulations and pre-visit veterinary checklists as defined in the study protocol (e.g., vaccination status, parasite control, and regular veterinary follow-up).
  * Patient agitation, defined as a Richmond Agitation-Sedation Scale (RASS) score > 0 (monitored every 4 hours per standard practice), before or during the visit.
  * Any other reason preventing the animal from entering the ICU or the patient's room before or during the visit (including patient discharge from ICU before the visit could be scheduled).
Pre-visit ICU staff satisfaction-related survey | Immediately before the intervention
  Pre-visit survey of ICU staff (including all clinical and non-clinical personnel such as physicians, nurses, therapists, hygiene and cleaning staff, administrative assistants, and supervisors) to assess their opinions and any potential concerns regarding the visit.
Post-visit ICU staff satisfaction-related survey | Immediately after the intervention
  Post-visit survey of the same ICU staff to assess their opinion and level of satisfaction.
Post-visit satisfaction survey of the patient's relative(s) who accompanied the dog | Immediately after the intervention
Patient satisfaction survey | ICU discharge (within a maximum of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Jabaudon, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No